CLINICAL TRIAL: NCT00814411
Title: A Randomized Trial of Group vs. Individual Family Planning Counseling in Ghana
Brief Title: A Trial of Group Versus Individual Family Planning Counseling in Ghana
Acronym: GCFP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Kwame Nkrumah University of Science and Technology (Other)
Responsible Party: Hilary Schwandt, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GCFP
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Last update posted 2008-12-24 (Estimated); Status verified 2008-12

CONDITIONS: Contraception
Keywords: contraception; noninferiority; intention; family planning counseling; post abortion care; Family planning intention among women with unmet need

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Counseling (Experimental): Group family planning counseling
  Interventions: Behavioral: group family planning counseling
- Individual Counseling (Active Comparator): Individual family planning counseling with gynecological patients who have unmet need
  Interventions: Behavioral: Individual family planning counseling

INTERVENTIONS:
Behavioral: group family planning counseling — group family planning counseling for gynecological patients with unmet need
  Arms: Group Counseling
Behavioral: Individual family planning counseling — Individual family planning counseling with gynecological patients - the current standard of care
  Arms: Individual Counseling

SUMMARY:
This study uses a randomized, noninferiority design to determine whether group family planning counseling is as effective as individual family planning counseling among gynecological patients with unmet need at two teaching hospitals in Ghana.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* fertile
* desires to delay pregnancy for at least 12 months

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Contraceptive Intention | Follow-up

SECONDARY OUTCOMES:
Modern contraceptive method knowledge | baseline and follow-up

CONTACTS AND LOCATIONS:
Locations (3):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States
- Ghana (2):
  - Komfo Anokye Teaching Hospital, Kumasi, Ashanti Region
  - Korle Bu Teaching Hospital, Accra, Greater Accra Region